CLINICAL TRIAL: NCT04350281
Title: An Open-label Randomized Controlled Trial on Interferon β-1b and Hydroxychloroquine Combination Versus Hydroxychloroquine Alone, as Treatment for COVID-19 Infection
Brief Title: Double Therapy With IFN-beta 1b and Hydroxychloroquine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ivan FN Hung MD, Professor of Medicine, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 20-211
Record Dates: First submitted 2020-04-13; First posted 2020-04-17 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: COVID
Keywords: IFN-beta 1b; hydroxychloroquine; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Interferon beta-1b; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): Subcutaneous injection of interferon β-1b 1mL (0.25mg; 8 million IU) consecutively on day 1 to day 3 and hydroxychloroquine 800mg on day 1, then 400mg daily for 2 days plus standard care
  Interventions: Drug: Interferon Beta-1B; Drug: Hydroxychloroquine
- Control group (Active Comparator): Hydroxychloroquine 800mg on day 1, then 400mg daily for 2 days plus standard care alone.
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Interferon Beta-1B — Daily subcutaneous injection of interferon β-1b 1mL (0.25mg; 8 million IU) consecutively on day 1 to day 3
  Arms: Treatment group
Drug: Hydroxychloroquine — Hydroxychloroquine 800mg on day 1, then 400mg daily for 2 days

SUMMARY:
The novel coronavirus (SARS-CoV-2), is a single-stranded RNA coronavirus. The virus was first isolated from patients presented with pneumonia in Wuhan in December 2019. Sequences of the Wuhan betacoronavirus show similarities to betacoronaviruses found in bats, sharing a common ancestor with the 2003 SARS coronavirus (SARS-CoV) and the bat coronavirus HKU9, a virus found in fruit bats. Similar to SARS-CoV, it is a member of Beta-CoV lineage B. Five genomes of the novel coronavirus have been initially isolated and reported including BetaCoV/Wuhan/IVDC-HB-01/2019, BetaCoV/Wuhan/IVDC-HB-04/2020, BetaCoV/Wuhan/IVDC-HB-05/2019, BetaCoV/Wuhan/WIV04/2019, and BetaCoV/Wuhan/IPBCAMS-WH-01/2019 from the China CDC.

The SARS-CoV-2 has since spread from China to the rest of the world. As of 5 April 2020, more than 1.05 million people been confirmed to have infected by SARS-CoV-2, resulting in more than 500,000 deaths. No specific antiviral treatment for the SARS-CoV-2 is currently available, but existing medication could be repurposed.

Genetic sequencing demonstrated similarity of the SARS-CoV-2 to the SARS-CoV and MERS CoV.2 We expect patients infected with the SARS-CoV-2 will also present similarly with initial upper respiratory tract symptoms including fever, cough, sputum, myalgia and shortness or breath. More severe cases might complicate with pneumonia and required ventilatory or ECMO support. According to our previous studies in 2003 on patients hospitalized for severe SARS-CoV, the viral load peaked between day 7 from symptoms onset and coincided with clinical deterioration of pneumonia and respiratory failure, with majority of the patients required intensive care support. Higher viral load isolated from different human system also correlated with worsened SARS manifestation and complications.

Previously, the investigators have demonstrated that interferon-beta 1b, commonly used in the treatment of multiple sclerosis and lopinavir/ ritonavir, also demonstrated to improve the outcome of MERS-CoV infection in a non-human primate model of common marmoset.

A non-randomized trial has also suggested that a combination of hydroxychloroquine and azithromycin might be effective in suppressing SARS-CoV-2 viral load in patients, despite in-vitro activity was only found in hydroxychloroquine.

Therefore, the investigators propose to conduct an open-label randomized controlled trial on a short course of interferon β-1b and hydroxychloroquine combination treatment for patients hospitalized for COVID-19 infection.

DETAILED DESCRIPTION:
This is a prospective open-label randomised controlled trial among adult patients hospitalised after April 2020 for virologically confirmed SARS-CoV-2 infection.

Patients will be randomly assigned to either the treatment group: a 3-day course of 3 doses of subcutaneous injection of interferon β-1b 1mL (0.25mg; 8 million IU) consecutively on day 1 to day 3 and hydroxychloroquine 800mg on day 1, then 400mg daily for 2 days plus standard care, or the control group: a 3-day course of hydroxycholoroquine 800mg on day 1, then 400mg daily for 2 days plus standard care alone (1:1).

For the control group, if the day 4 nasopharyngeal swab (NPS) viral load remains positive, then patients will receive another 3 days of subcutaneous injection of interferon β-1b 1mL (0.25mg; 8 million IU) and hydroxychloroquine 400mg daily.

ELIGIBILITY:
Inclusion Criteria:

1. Recruited subjects include all adult patients ≥18 years hospitalized for virologic confirmed SARS-CoV-2 infection.
2. All subjects give written informed consent. For patients who are critically ill, requiring ICU, ventilation or confused, informed consent will be obtained from spouse, next-of-kin or legal guardians.
3. Subjects must be available to complete the study and comply with study procedures. Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

1. Inability to comprehend and to follow all required study procedures.
2. Allergy or severe reactions to the study drugs
3. Patients with known prolonged QTc syndrome, ventricular cardiac arrhythmias, including torsade de pointes, second or third degree heart block, QTc interval >480ms
4. Patients taking medication that will potentially interact with l interferon beta-1b or hydroxychloroquine
5. Patients with known underlying retinopathy
6. Patients with G6PD deficiency
7. Patients with known history of severe depression
8. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to recruitment in this study or expect to receive an experimental agent during this study.
9. To participate in an unrelated trial during the current clinical trial. Nevertheless, the patients have the right to withdraw from the current clinical trial to join another clinical trial.
10. Have a history of alcohol or drug abuse in the last 5 years.
11. Have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Time to negative NPS viral load | 4 weeks
  Time to negative NPS SARS-CoV-2 viral RT-PCR

SECONDARY OUTCOMES:
Time to NEWS 0 | 4 weeks
  Time to complete allevation of symptoms as defined by NEWS of 0 maintained for 24 hours
Length of Hospitalisation | 4 weeks
  Days of hospital stay
Time to negative viral load in all clinical samples | 4 weeks
  Time to negative SARS-CoV-2 viral RT-PCR in all clinical samples
Adverse events | 4 weeks
  Treatment related adverse events
Mortality | 30 days
  30-day mortality
Inflammatory markers changes | 4 weeks from diagnosis
  Cytokine/ chemokine

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN Hung, MD FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No